CLINICAL TRIAL: NCT04027998
Title: Median Nerve Strain and Applied Pressure Measurement in the Carpal Tunnel Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Yuichi Yoshii, Associate Professor, Department of Orthopaedic Surgery, Tokyo Medical University
Other Study IDs: 14-5
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carpal tunnel syndrome: group of carpal tunnel syndrome patients
  Interventions: Diagnostic Test: strain and applied pressure measurement
- Control group: group of healthy controls
  Interventions: Diagnostic Test: strain and applied pressure measurement

INTERVENTIONS:
Diagnostic Test: strain and applied pressure measurement — Measurement of median nerve strain and applied pressure at proximal carpal tunnel level

SUMMARY:
The aim of this study is to investigate diagnostic accuracy of median nerve strain and applied pressure measurement . Idiopathic carpal tunnel syndrome patients and healthy controls will be evaluated by ultrasound. Median nerve strain, pressure applied to the skin will be measured at the proximal part of the carpal tunnel. The parameters will be compared between patients and controls, and before and after the open carpal tunnel release in the patients.

DETAILED DESCRIPTION:
The aim of this study is to investigate diagnostic accuracy of median nerve strain and applied pressure measurement . Idiopathic carpal tunnel syndrome patients and healthy controls will be evaluated by ultrasound. Median nerve strain, pressure applied to the skin, and ratio of pressure-strain will be measured at the proximal part of the carpal tunnel. In addition, distal latencies in the motor and sensory nerve conductions studies and cross-sectional area of median nerve will be measured. The parameters will be compared between patients and controls, and before and after the open carpal tunnel release in the patients.

ELIGIBILITY:
Inclusion Criteria:

* carpal tunnel syndrome patients and asymptomatic control

Exclusion Criteria:

* Patients were excluded if there was a history of cervical radiculopathy, rheumatoid arthritis, gout, hemodialysis, sarcoidosis, amyloidosis, or traumatic injuries to the arm. Written consent was obtained from all study participants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: carpal tunnel syndrome patients and asymptomatic control
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04-03 (Actual); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
median nerve strain | through study completion, an average of 1 year
  Change of the median nerve strain from the initial measurement at 3, 6, 12 months after the treatment
applied pressure | through study completion, an average of 1 year
  Change of the applied pressure from the inital measurement at 3, 6, 12months after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuichi Yoshii, Principal Investigator — Tokyo Medical University Ibaraki Medical Center
Locations (1):
- Tokyo Medical University Ibaraki Medical Center, Ami, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoshii Y, Tung WL, Yuine H, Ishii T. Postoperative diagnostic potentials of median nerve strain and applied pressure measurement after carpal tunnel release. BMC Musculoskelet Disord. 2020 Jan 11;21(1):22. doi: 10.1186/s12891-019-3033-y. PMID 31926552